CLINICAL TRIAL: NCT00351078
Title: A Phase 2b Extension Study of PTC124 as an Oral Treatment for Nonsense-Mutation-Mediated Cystic Fibrosis
Brief Title: PTC124 for the Treatment of Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-005e-CF
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Nonsense mutation; Premature stop codon; CF; PTC124
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTC124 PO (Experimental): 4-, 4-, and 8-mg/kg TID first 14 days of cycle 10-, 10-, and 20-mg/kg TID second 14 days of cycle 28 day study
  Interventions: Drug: PTC124

INTERVENTIONS:
Drug: PTC124 — 4-,4-, and 8-mg/kg PO first 14 days 10-, 10-, and 20-mg/kg TID second 14 days

SUMMARY:
In some patients with cystic fibrosis (CF), the disease is caused by a nonsense mutation (premature stop codon) in the gene that makes the cystic fibrosis transmembrane regulator (CFTR) protein. PTC124 has been shown to partially restore CFTR production in animals with CF due to a nonsense mutation. In an ongoing Phase 2a study being performed at the Hadassah University Hospital - Mount Scopus in Israel, patients with nonsense-mutation-mediated CF have received PTC124 in two 14-day treatment courses. Preliminary results from that study indicate that PTC124 has pharmacodynamic activity of PTC124 in CF and that PTC124 can be safely administered in this patient population. This Phase 2b extension study is designed to evaluate the activity and safety of 3 months (approximately 84 days) of continuous treatment with PTC124 in the same patients who were enrolled to the Phase 2a study. The main purpose of this study is to understand whether PTC124 can be safely administered and achieve pharmacodynamic activity in patients with CF due to a nonsense mutation.

DETAILED DESCRIPTION:
In this study, the same patients who were enrolled in a previous study of PTC124 (protocol number PTC124-GD-005-CF) will be treated with the investigational drug PTC124 for a period of 84 days. Evaluation procedures (history, physical examination, blood and urine tests to assess organ function, electrocardiogram (ECG), chest x-ray, and CF-specific tests) to determine if a patient qualifies for the study will be performed within 21 days prior to the start of treatment. Eligible patients who elect to enroll in the study will be assigned to receive PTC124 treatment (based upon TEPD results from the previous study) at 1 of the 2 following dose levels:

* PTC124, given 3 times per day (TID) with a regimen of 4 mg/kg at breakfast, 4 mg/kg at lunch, and 8 mg/kg at dinner, or
* PTC124, given 3 times per day (TID) with a regimen of 10 mg/kg at breakfast, 10 mg/kg at lunch and 20 mg/kg at dinner.

During the study, PTC124 efficacy, safety, and pharmacokinetics will be evaluated periodically with measurement of transepithelial potential difference (TEPD), medical history, physical examinations, blood tests, urinalysis, sputum tests, ECGs, chest x-ray, and pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following conditions to be eligible for enrollment into the study:

* Completion of ≥ 1 cycle of PTC124 treatment in the previous Phase 2a study protocol (Protocol Number PTC124-GD-005-CF).
* Abnormal nasal epithelial TEPD total chloride conductance (a more electrically negative value than -5 mV for Δchloride-free+isoproterenol).
* FEV1 ≥ 40% of predicted for age, gender, and height.
* Oxygen saturation (as measured by pulse oximetry) ≥92% on room air.
* Willingness of male and female patients, if not surgically sterile, to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and follow-up periods.
* Negative pregnancy test (for females of childbearing potential).
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, and study restrictions.
* Ability to provide written informed consent.
* Evidence of signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

The presence of any of the following conditions will exclude a patient from enrollment in the study:

* Prior or ongoing medical condition, medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the patient, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.
* Ongoing acute illness including acute upper or lower respiratory infections within 2 weeks before start of study treatment in this study.
* History of major complications of lung disease (including recent massive hemoptysis or pneumothorax) within 2 months prior to start of study treatment in this study.
* Abnormalities on screening chest x-ray suggesting clinically significant active pulmonary disease other than CF, or new, significant abnormalities such as atelectasis or pleural effusion which may be indicative of clinically significant active pulmonary involvement secondary to CF.
* Hemoglobin <10 g/dL.
* Serum albumin <2.5 g/dL.
* Abnormal liver function (serum total bilirubin > the upper limit of normal, or serum ALT, AST, or GGT >2.0 times the upper limit of normal). Abnormal renal function (serum creatinine >1.5 times upper limit of normal).
* Pregnancy or breast-feeding.
* History of solid organ or hematological transplantation.
* Exposure to another investigational drug within 14 days prior to start of study treatment in this study.
* Ongoing participation in any other therapeutic clinical trial.
* Ongoing use of thiazolidinedione peroxisome proliferator-activated receptor gamma (PPAR γ) agonists, eg, rosiglitazone (Avandia® or equivalent) or pioglitazone (Actos® or equivalent).
* Change in intranasal medications (including use of corticosteroids, cromolyn, ipratropium bromide, phenylephrine, or oxymetazoline) within 7 days prior to start of study treatment in this study.
* Change in treatment with systemic or inhaled corticosteroids within 7 days prior to start of study treatment in this study.
* Use of or requirement for inhaled gentamicin or amikacin within 14 days prior to start of study treatment in this study or during study treatment.
* Requirement for systemic aminoglycoside antibiotics within 14 days prior to start of study treatment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
CFTR activity as assessed by nasal transepithelial potential difference (TEPD) | 84 days

SECONDARY OUTCOMES:
Side effects | 84 days
Presence of CFTR protein and mRNA | 84 days
Compliance with treatment | 84 days
Lung function | 84 days
Sputum test | 84 days
PTC124 pharmacokinetics | 84 days'
Changes in CF symptoms | 84 days
Changes in weight | 84 days
Changes in cough | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Kerem, MD, Principal Investigator — Hadassah University Hospital - Mount Scopus
Locations (1):
- Hadassah University Hospital - Mount Scopus, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilschanski M, Miller LL, Shoseyov D, Blau H, Rivlin J, Aviram M, Cohen M, Armoni S, Yaakov Y, Pugatsch T, Cohen-Cymberknoh M, Miller NL, Reha A, Northcutt VJ, Hirawat S, Donnelly K, Elfring GL, Ajayi T, Kerem E. Chronic ataluren (PTC124) treatment of nonsense mutation cystic fibrosis. Eur Respir J. 2011 Jul;38(1):59-69. doi: 10.1183/09031936.00120910. Epub 2011 Jan 13. PMID 21233271
- See also: Provides description of the PTC124 study from which the patients will be enrolled into this study. — http://clinicaltrials.gov/ct/show/NCT00237380?order=2